CLINICAL TRIAL: NCT00922779
Title: Safety and Tolerability of Ribavirin (RO 20-9963) in Combination With Peginterferon Alfa-2a (40 kD)in Patients With Chronic Hepatitis C
Brief Title: A Study of Ribavirin in Combination With PEGASYS (Peginterferon Alfa-2a (40KD))in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16709
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180micrograms sc weekly for 12-48 weeks
Drug: ribavirin — 800mg, or 1000-1200mg, po daily (dependent on HCV genotype and body weight)

SUMMARY:
This single arm study will evaluate the safety and tolerability of ribavirin in combination with PEGASYS in patients with chronic hepatitis C. Patients will receive ribavirin 800mg, or 1000-1200mg po daily, according to HCV genotype and body weight (< and >75kg)in combination with PEGASYS 180micrograms sc weekly. The anticipated time on study treatment is 3-12 months, and the target sample size is >500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* serological evidence of chronic hepatitis C;
* detectable serum HCV-RNA;
* liver biopsy findings consistent with a diagnosis of chronic hepatitis C.

Exclusion Criteria:

* history or other evidence of a medical condition associated with chronic liver disease other than HCV;
* co-infection with active hepatitis A or B;
* hepatocellular carcinoma;
* patients with severe cardiovascular disease whose condition may worsen due to acute anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6661 (Actual)
Dates: Start 2002-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- Russia (42):
  - Arkhangelsk
  - Barnaul
  - Blagoveshchensk
  - Cheboksary
  - Chelyabinsk
  - Cherepovets
  - Chita
  - Irkutsk
  - Izhevsk
  - Kazan'
  - Kemerovo
  - Khabarovsk
  - Kirov
  - Krasnodar
  - Krasnoyarsk
  - Lipetsk
  - Makhachkala
  - Moscow
  - Nizhny Novgorod
  - Novokuznetsk
  - Novosibirsk
  - Novoural'sk
  - Omsk
  - Orenburg
  - Petropavlovsk-Kamchatskiy
  - Rostov-on-Don
  - Saint Petersburg
  - Salekhard
  - Samara
  - Saratov
  - Sashi
  - Stavropol
  - Surgut
  - Tomsk
  - Tyumen
  - Ufa
  - Ulan-Ude
  - Vladivostok
  - Volgograd
  - Yakutsk
  - Yekaterinburg
  - Yujno-sakhalinsk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7799 participants were screened, of which 6661 participants were included in the study.
Groups:
- Ribavirin + Peginterferon Alfa-2a: Participants with genotype 1 received ribavirin oral tablets daily depending on the body weight. Participants with body weight of less than 75 kilograms (kg) received dose of 400 milligrams (mg) (2 tablets of 200 mg) in morning and 600 mg (3 tablets of 200 mg) in evening, and participants with body weight of 75 kg or more, received dose of 600 mg (3 tablets of 200 mg) in the morning and evening along with Peginterferon (PEG-INF) Alfa-2a 180 micrograms per milliliter (µg/mL) subcutaneous (SC) injection once weekly for 12 to 48 weeks. Participants with other genotypes received ribavirin dose of 400 mg (2 tablets of 200 mg) in morning and evening along with PEG-INF Alfa-2a 180 µg/mL SC injection once weekly for 12 to 24 weeks.
Period: Overall Study
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Started | 6661
Completed | 4334
Not Completed | 2327
Not completed — Adverse Event | 67
Not completed — Pregnancy | 7
Not completed — Withdrawal by Subject | 308
Not completed — Lost to Follow-up | 44
Not completed — Other | 27
Not completed — Missing | 1874

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Groups:
- Ribavirin + Peginterferon Alfa-2a: Participants with genotype 1 received ribavirin oral tablets daily depending on the body weight. Participants with body weight of less than 75 kg received dose of 400 mg (2 tablets of 200 mg) in morning and 600 mg (3 tablets of 200 mg) in evening, and participants with body weight of 75 kg or more, received dose of 600 mg (3 tablets of 200 mg) in the morning and evening along with PEG-INF Alfa-2a 180 µg/mL SC injection once weekly for 12 to 48 weeks. Participants with other genotypes received ribavirin dose of 400 mg (2 tablets of 200 mg) in morning and evening along with PEG-INF Alfa-2a 180 µg/mL SC injection once weekly for 12 to 24 weeks.
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Number analyzed (Participants) | 6661
Age, Continuous [Mean (Standard Deviation); unit: Years] — Here, number of participants analyzed for baseline measure "age" was 6622.
  Years | 34.21 (9.81)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 4396
  Female | 2250
  Missing | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with non-serious AEs were exclusive of serious AEs.
Time Frame: From signing of informed consent up to end of study (up to Week 72)
Population: Safety analysis population included all participants who received at least one therapeutic dose of ribavirin.
Measure: Number; unit: Participants
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Number analyzed (Participants) | 6661
Participants
  Non Serious AEs | 2058
  SAEs | 67

2. Secondary Outcome: Percentage of Participants With Sustained Virological Response (SVR) at 24 Weeks After End of Therapy
Description: SVR at 24 weeks after end of therapy was defined as a negative result of HCV Ribonucleic Acid (HCV RNA) qualitative assay 24 weeks after end of therapy. Percentage of participants with SVR was calculated as [number of participants with negative results of HCV RNA qualitative assay 24 weeks after end of therapy divided by the total number of participants analyzed] multiplied by 100. The participants who failed to undergo tests at 24 weeks after completion of therapy were considered not amenable to therapy.
Time Frame: 24 weeks after end of therapy (Week 72)
Population: Intent-to-treat (ITT) population included all participants who received at least one therapeutic dose of ribavirin.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Number analyzed (Participants) | 6661
Percentage of Participants | 50.9

3. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA at Weeks 12, 24 and 48 After Therapy Initiation
Description: HCV RNA levels of < 50 International Units per milliliter (IU/mL) were defined as undetectable HCV RNA. The percentage of participants with undetectable HCV RNA was calculated as [number of participants with undetectable HCV RNA divided by the total number of participants analyzed] multiplied by 100 for Weeks 12, 24 and 48.
Time Frame: Weeks 12,24 and 48 After Therapy Initiation
Population: ITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Number analyzed (Participants) | 6661
Percentage of Participants
  Week 12 | 58.8
  Week 24 | 69.7
  Week 48 | 24.8

4. Secondary Outcome: Percentage of Participants With Change in Hemoglobin Level
Description: Change in hemoglobin level (compared to baseline) was reported as "significant decrease", "Normal" (no change), "Increase", "Decrease", and "Missing". Significant decrease was defined as per Investigator's discretion.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 48 and follow-up Weeks 4 (Week 52), 12 (Week 60), and 24 (Week 72)
Population: ITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Number analyzed (Participants) | 6661
Percentage of Participants
  Week 2, Significant decrease | 13.5
  Week 2, Normal | 32.4
  Week 2, Increase | 11.7
  Week 2, Decrease | 32.3
  Week 2, Missing | 10.0
  Week 4, Significant decrease | 27.9
  Week 4, Normal | 21.0
  Week 4, Increase | 6.9
  Week 4, Decrease | 35.1
  Week 4, Missing | 9.1
  Week 8, Significant decrease | 35.4
  Week 8, Normal | 15.3
  Week 8, Increase | 5.1
  Week 8, Decrease | 31.5
  Week 8, Missing | 12.8
  Week 12, Significant decrease | 38.9
  Week 12, Normal | 15.2
  Week 12, Increase | 4.7
  Week 12, Decrease | 30.1
  Week 12, Missing | 11.1
  Week 24, Significant decrease | 34.9
  Week 24, Normal | 13.6
  Week 24, Increase | 4.6
  Week 24, Decrease | 25.4
  Week 24, Missing | 21.5
  Week 36, Significant decrease | 16.2
  Week 36, Normal | 4.1
  Week 36, Increase | 1.7
  Week 36, Decrease | 9.1
  Week 36, Missing | 69.0
  Week 48, Significant decrease | 13.7
  Week 48, Normal | 3.8
  Week 48, Increase | 1.7
  Week 48, Decrease | 7.7
  Week 48, Missing | 73.1
  Follow-up Week 4, Significant decrease | 11.5
  Follow-up Week 4, Normal | 18.5
  Follow-up Week 4, Increase | 6.8
  Follow-up Week 4, Decrease | 19.6
  Follow-up Week 4, Missing | 43.7
  Follow-up Week 12, Significant decrease | 5.8
  Follow-up Week 12, Normal | 23.0
  Follow-up Week 12, Increase | 10.2
  Follow-up Week 12, Decrease | 16.1
  Follow-up Week 12, Missing | 44.8
  Follow-up Week 24, Significant decrease | 4.7
  Follow-up Week 24, Normal | 27.5
  Follow-up Week 24, Increase | 12.2
  Follow-up Week 24, Decrease | 15.5
  Follow-up Week 24, Missing | 40.2

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to end of study (up to Week 72)
Arm/Group | Ribavirin + Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 67/6661
Other Adverse Events (participants affected / at risk) | 1674/6661
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin + Peginterferon Alfa-2a (N=6661)
Pyelonephritis acute (Infections and infestations) | 2
Acute tonsillitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Chronic hepatitis C (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Hepatitis G (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Cardiovascular insufficiency (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Completed suicide (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Delusional disorder, persecutory type (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Cranial nerve disorder (Nervous system disorders) | 1
IIIrd nerve disorder (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Injury (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Macular oedema (Eye disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Chronic tonsillitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin + Peginterferon Alfa-2a (N=6661)
Asthenia (General disorders) | 905
Influenza like illness (General disorders) | 833
Pyrexia (General disorders) | 371
Anaemia (Blood and lymphatic system disorders) | 459
Weight loss poor (Metabolism and nutrition disorders) | 343

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.